CLINICAL TRIAL: NCT05840393
Title: The Effect of Roy Adaptation Model-Based Discharge Training on Quality of Life and Adaptation of Palliative Care Patients and Caregivers
Brief Title: The Effect of Discharge Education Based on Roy Adaptation Model on Palliative Care Patients and Caregivers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, ELİF TUĞBA UYGUN, Principal Investigator Phd candidate of nursing, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EUYGUN
Record Dates: First submitted 2023-03-29; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Nurse's Role; Nutritional Deficiency; Adaptation Reaction
Keywords: Discharge training; Nutrition; Quality of life; Adaptation; Palliative care
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Discharge training based on the Roy adaptation model (Experimental): Oncologic palliative care patients and caregivers in this group will receive discharge training based on the Roy adaptation model.
  Interventions: Other: Discharge training based on Roy adaptation model
- Control Group: Standard discharge training (No Intervention): Oncologic palliative care patients and caregivers in this group will not receive any training other than the discharge training routinely applied in the clinic.

INTERVENTIONS:
Other: Discharge training based on Roy adaptation model — The Roy Adaptation Model consists of four main areas of adaptation. In this study, the content of the discharge education given within the scope of the adaptation areas of the Roy Adaptation Model will be continued with information such as home nutrition process, pain, anxiety, fear, stress and coping methods, addressing changing roles and responsibilities, communication, problem solving and utilizing social support. A booklet will be prepared to increase the effectiveness of discharge training based on the Roy Adaptation Model and the booklet will be used as a guide in the training program.
  Arms: Intervention Group: Discharge training based on the Roy adaptation model

SUMMARY:
This research will be carried out in order to reveal how the discharge education that will be formed in line with the Roy Adaptation Model for oncological palliative care patients and caregivers will affect the nutritional outcomes, quality of life and adaptation difficulties of the patients, coping and adaptation processes of caregivers, their quality of life and their level of knowledge about nutritional care.

DETAILED DESCRIPTION:
Today, with the improvement of living conditions and the development of technology in the field of medicine, life expectancy and the elderly population are increasing every day. This situation leads to an increase in the number of individuals with chronic diseases and increases the need for palliative care services day by day.

In palliative care; meeting the needs of patients, families and caregivers, ensuring an increase in the quality of life by supporting patients physically, psychologically, socially and spiritually in the last period of their lives, and providing care according to the needs of the individual and family / caregivers in the process of death and mourning. Patients in need of palliative care face many problems such as pain, nausea, vomiting, fatigue, depression, dyspnea, dehydration, constipation, weakness, fatigue, delirium, disorientation and malnutrition that develop due to the disease and reduce the quality of life. In the care of palliative patients, caregivers play an important role in symptom control and helping the patient to maintain life activities, especially nutrition.İnforming healthy/patient individuals and their families/caregivers about healthy lifestyle changes is within the scope of the nurse's educational and counseling roles. In the palliative care process, it is stated that the lack of discharge training on nutrition may lead to significant problems.Nurses need to benefit from theories and models while applying qualified nursing care to the individual, family or community, managing the health of the people to whom they apply nursing care, supporting them to adapt to the new process they live in, and explaining the data they obtain in a scientific sense.

In this direction, in this study, the effect of the discharge training to be created in line with the Roy Adaptation Model, one of the nursing models, on oncological palliative care patients with malnutrition and receiving nutritional support and their caregivers will be revealed.

This research will be conducted in a prospective, randomized experimental design with pretest-posttest experimental and control groups. The sample size of the study will consist of oncological palliative care patients and caregivers who meet the inclusion criteria and agree to participate in the study. The patients and caregivers to be included in the sample of the study will be randomly divided into two groups as experimental and control groups.

The sample size of the study was calculated by power analysis. The power of the study was determined as 42 oncological palliative care patients and caregivers (minimum n=21 patients and caregivers for each group) as a result of the analysis performed according to the data of a referenced study (taking the effect size as 0.9, 80% power value and 0.05% margin of error and confidence interval). In order to increase the reliability of the study and to be able to apply parametric tests, the total sample size was determined as n:60, including 30 oncological palliative care patients and caregivers of the experimental group and 30 oncological palliative care patients and caregivers of the control group, taking into account data losses (dropout from the study, death, etc.). Randomization in the study will be provided by using the randomization method in simple random order. Patients were randomly selected to the experimental and control groups. The data will be evaluated with the SPSS (Statistical Package of SocialSciences) 24.0 package program.

Data; Descriptive Information Form Specific to Oncologic Palliative Care Patients, Nutritional Risk Screening Test-2002 (NRS-2002), EORTC QLQ-C30 Quality of Life Scale, Scale for Assessing Difficulties of Adaptation in the Elderly, Nutritional Follow-up Form, Telephone Counseling Follow-up Form, Descriptive Information Form Specific to Caregivers of Oncologic Palliative Care Patients, Coping and Adaptation Process Scale, World Health Organization Quality of Life Scale (WHOQOL-BREF-TR), Information Form Including Opinions on Nutritional Care will be collected.

ELIGIBILITY:
Inclusion Criteria:

* 65 years of age or older,
* Receiving inpatient treatment in a palliative care clinic for an existing oncological disease,
* To be discharged home after the end of palliative care treatment,
* Continuing home nutritional support (Percutaneous Endoscopic Gastrostomy/PEG) during hospitalization and after discharge,
* NRS-2002 malnutrition risk score of 3 and above during hospitalization (data to be obtained from the patient file),
* To have the ability to understand and speak Turkish,
* To be able to communicate by phone,
* No disability in terms of state of consciousness and sensory organs,
* Volunteering to participate in the research.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria, patients who die or whose condition worsens during the research process, and patients who do not volunteer to participate in the research and their caregivers will be excluded from the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Quality of Life Scale | Pre-discharge and 3-month post-discharge follow-up of the patients
  The quality of life of palliative care patients will be assessed using the EORTC QLQ-C30 Quality of Life Scale (consisting of 30 items, the first 28 of which are four-point Likert-type scales and the items are None: 1, Somewhat: 2, Somewhat: 3 or Very: 4 points. Question 29 asks the patient to rate their health on a scale from 1 to 7 (1: Very poor and 7: Excellent) and question 30 asks the patient to rate their overall quality of life. High scores in this section indicate a high quality of life and low scores indicate a low quality of life.) The World Health Organization Quality of Life Scale (It consists of 26 questions related to physical, mental, environmental, social relations and general health status. Each domain is calculated over 20 points or 100 points. A high score indicates a high quality of life).
Compliance Scale | Pre-discharge and 3-month post-discharge follow-up of the patients
  The adaptation of palliative care patients will be determined using the Difficulty of Adaptation in the Elderly Assessment Scale (a four-point Likert-type scale consisting of 24 items, scored as "not at all, a little, quite, a lot"). As the score obtained from the scale increases, the level of adaptation to old age decreases.
  The adaptation of caregivers will be determined using the Coping and Adaptation Process Scale. The scale, which is based on the Roy Adaptation Model and the concepts related to the cognitive process it defines and used to determine the coping and adaptation strategies of individuals in critical and difficult situations, is a four-point Likert-type scale consisting of five sub-dimensions and 47 items (each statement is answered "never, rarely, sometimes, always"). As the scores obtained from the scale increase, it is evaluated as the use of effective coping methods and adaptation increases.

CONTACTS AND LOCATIONS:
Overall Officials: Aylin ÖZAKGÜL, Study Director — Istanbul University - Cerrahpasa

REFERENCES:
- [Background] Adelman RD, Tmanova LL, Delgado D, Dion S, Lachs MS. Caregiver burden: a clinical review. JAMA. 2014 Mar 12;311(10):1052-60. doi: 10.1001/jama.2014.304. PMID 24618967
- [Background] Fitch MI, Fliedner MC, O'Connor M. Nursing perspectives on palliative care 2015. Ann Palliat Med. 2015 Jul;4(3):150-5. doi: 10.3978/j.issn.2224-5820.2015.07.04. PMID 26231811
- [Background] Stajduhar KI, Funk L, Cohen SR, Williams A, Bidgood D, Allan D, Norgrove L, Heyland D. Bereaved family members' assessments of the quality of end-of-life care: what is important? J Palliat Care. 2011 Winter;27(4):261-9. PMID 22372280
- [Background] Starke J, Schneider H, Alteheld B, Stehle P, Meier R. Short-term individual nutritional care as part of routine clinical setting improves outcome and quality of life in malnourished medical patients. Clin Nutr. 2011 Apr;30(2):194-201. doi: 10.1016/j.clnu.2010.07.021. PMID 20937544
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Barker LA, Gout BS, Crowe TC. Hospital malnutrition: prevalence, identification and impact on patients and the healthcare system. Int J Environ Res Public Health. 2011 Feb;8(2):514-27. doi: 10.3390/ijerph8020514. Epub 2011 Feb 16. PMID 21556200
- [Background] Burgos R, Sarto B, Elio I, Planas M, Forga M, Canton A, Trallero R, Munoz MJ, Perez D, Bonada A, Salo E, Lecha M, Enrich G, Salas-Salvado J; Group for the Study of Malnutrition in Hospitals in Catalonia. Prevalence of malnutrition and its etiological factors in hospitals. Nutr Hosp. 2012 Mar-Apr;27(2):469-76. doi: 10.1590/S0212-16112012000200018. PMID 22732970
- [Background] Elia M. Defining, Recognizing, and Reporting Malnutrition. Int J Low Extrem Wounds. 2017 Dec;16(4):230-237. doi: 10.1177/1534734617733902. Epub 2017 Nov 16. PMID 29145755
- [Background] Yoder LH. Using the Roy adaptation model: a program of research in a Military Nursing Research Service. Nurs Sci Q. 2005 Oct;18(4):321-3; discussion 320. doi: 10.1177/0894318405280382. No abstract available. PMID 16294464
- [Background] Guzelant A, Goksel T, Ozkok S, Tasbakan S, Aysan T, Bottomley A. The European Organization for Research and Treatment of Cancer QLQ-C30: an examination into the cultural validity and reliability of the Turkish version of the EORTC QLQ-C30. Eur J Cancer Care (Engl). 2004 May;13(2):135-44. doi: 10.1111/j.1365-2354.2003.00435.x. PMID 15115469
- [Background] Kaya A, Boz I. The development of the Professional Values Model in Nursing. Nurs Ethics. 2019 May;26(3):914-923. doi: 10.1177/0969733017730685. Epub 2017 Sep 20. PMID 28929939
- [Background] Kondrup J, Rasmussen HH, Hamberg O, Stanga Z; Ad Hoc ESPEN Working Group. Nutritional risk screening (NRS 2002): a new method based on an analysis of controlled clinical trials. Clin Nutr. 2003 Jun;22(3):321-36. doi: 10.1016/s0261-5614(02)00214-5. PMID 12765673
- [Background] Lopez-Contreras MJ, Torralba C, Zamora S, Perez-Llamas F. Nutrition and prevalence of undernutrition assessed by different diagnostic criteria in nursing homes for elderly people. J Hum Nutr Diet. 2012 Jun;25(3):239-46. doi: 10.1111/j.1365-277X.2012.01237.x. Epub 2012 Feb 23. PMID 22360373